CLINICAL TRIAL: NCT06888427
Title: Qualitative Analysis of Factors Affecting Perioperative Sleep Quality During Scheduled Surgery
Brief Title: Sleep Longitudinal Exploration of the Experience of Patients
Acronym: SLEEP
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24-PP-18
Record Dates: First submitted 2025-03-13; First posted 2025-03-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Sleep
Keywords: sleep, surgical intervention
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients requiring scheduled surgery with post-operative hospitalization: Patients will pass questionnaires to assess their postoperative sleep quality
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — With the help of a questionnaires, determination of postoperative sleep quality

SUMMARY:
Many epidemiological studies report that insomnia is common after fifty years in the general population but also in the post-operative period of surgery. Preoperatively, sleep quality can be disturbed by fear of general anesthesia and surgery. Postoperatively, it seems to be altered by pain, the ambient environment and night care.

Literature shows that the occurrence of post-operative sleep disorders seems to lead to (increased) hypnotic consumption in patients who did not consume them in the pre-operative phase with known risks of dependence.

Nowadays , general anesthesia is widely practiced worldwide. However, despite continuous improvement in techniques, a large number of patients still experience poor quality postoperative sleep, even with short-term anesthesia.

It therefore appears that general anesthesia disrupts the circadian rhythm of patients, even if the mechanisms are still poorly understood.

Thus, sleep deprivation could be responsible of physiological alterations that are still unknown, such as delayed healing or impaired respiratory muscle performance, promoting postoperative complications.

The aim of this study is to identify the factors impacting the quality of sleep of patients undergoing scheduled surgery during the first postoperative night. And its implication on the occurrence of drowsiness described by the patient the day after their surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18 years or older;
* Subject scheduled to undergo surgery under general anesthesia (orthopedic, thoracic, vascular or visceral surgery);
* Subject able to complete a self-administered questionnaire;
* Subject having given oral consent;

Exclusion Criteria:

* Subject wishing to discontinue participation in the study before the end;
* Subject for whom the surgical procedure could not be performed after admission to the operating room (whatever the reason);
* Subject for whom the surgical procedure was performed urgently before the date initially scheduled (whatever the reason);
* Subject for whom a serious perioperative complication occurred during the surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older thant 18 requiring scheduled surgery with post-operative hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-10-23 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of factors influencing sleep quality | Day 1 post-operative
  Sleep quality will be assessed using a self-questionnaire called Spiegel. It includes 3 items assessing sleep with a gradation from 0 to 5. An overall score is calculated, ranging from 0 (worst possible experience) to 15 (very good quality of sleep).

SECONDARY OUTCOMES:
Determination of Sleepiness | Day 1 post-operative
  The occurrence of drowsiness will be assessed using a single-choice question with 5 options (5: absence of drowsiness; 0 : presence of drowsiness)
Determination of patient's perioperative satisfaction | Day 1 post-operative
  The perioperative patient' satisfaction assessed by the EVAN questionnaire. This questionnaire contains 22 items allowing a global analysis of patient satisfaction (1-100 points)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Maurice - Szamburski, MD-PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: No